CLINICAL TRIAL: NCT06428253
Title: A Single Center, Subject & Evaluator-blind, Randomized, Matched Pairs, Active-controlled, Confirmatory Study to Evaluate the Efficacy and Safety of HMM1-022 in Temporary Correction of Crow's Feet
Brief Title: Efficacy and Safety of HMM1-022 in Temporary Correction of Crow's Feet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Humedix Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMM1-022
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Crow's Feet

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: subject/evaluator blinding
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HMM1-022 (Experimental): Participants will receive injections into the wrinkles at the corners of each eye, up to 1 mL each, four times at two-week intervals.
  Interventions: Device: HMM1-022
- REJURAN® (Active Comparator): Participants will receive injections into the wrinkles at the corners of each eye, up to 1 mL each, four times at two-week intervals.
  Interventions: Device: HMM1-022

INTERVENTIONS:
Device: HMM1-022 — intradermal injection

SUMMARY:
The purpose of this study is to compare the efficacy and safety of HMM1-022 with Rejuran to improve Crow's feet

DETAILED DESCRIPTION:
A single center, subject & evaluator-blind, randomized, matched pairs, active-controlled, confirmatory study to evaluate the efficacy and safety of HMM1-022 in temporary correction of Crow's feet

ELIGIBILITY:
Inclusion criteria

* Adult aged 19 years or older
* Individuals who have voluntarily decided to participate in the clinical trial after receiving and understanding a detailed explanation, and who have provided written consent
* Individuals who have agreed to discontinue all dermatological treatments, including wrinkle treatments around the eyes, during the clinical trial period

Exclusion criteria

1. Individuals with a history of anaphylaxis or severe allergic diseases that may affect the clinical trial
2. Individuals diagnosed with autoimmune diseases, sarcoid granulomatous pathology, or Osler's endocarditis
3. Individuals with hypersensitivity to the investigational medical device, its components (polynucleotide sodium, hyaluronic acid sodium, lidocaine), or other amide-type local anesthetics
4. Individuals with a history of bleeding disorders
5. Individuals with a history of facial nerve paralysis or ptosis
6. Individuals with significant facial asymmetry that may affect the clinical trial
7. Individuals with skin diseases, infections, or abnormalities such as scars in the eye area that could affect the clinical trial
8. Individuals with a history of keloid formation, hyperpigmentation, or hypertrophic scar in the evaluation area
9. Individuals with a history of malignant tumors within 5 years prior to Visit 1 (screening), except those with treated basal cell or squamous cell skin cancer not in the eye area, or treated cervical cancer
10. Individuals with clinically significant disorders or psychiatric conditions affecting the cardiovascular, gastrointestinal, respiratory, endocrine, immune, or central nervous systems, or those with conditions that may significantly impact the clinical trial
11. Individuals who have undergone or are scheduled to undergo treatments affecting the efficacy assessment of crow's feet wrinkles during the following periods:

    * Within 24 months before Visit 1 (screening) using Poly(L-Lactide) or Poly(ε-Caprolactone) for wrinkle treatment
    * Within 18 months before Visit 1 (screening) using Calcium hydroxylapatite (CaHA) for wrinkle treatment
    * Within 12 months before Visit 1 (screening) using hyaluronic acid for wrinkle treatment
    * Within 6 months before Visit 1 (screening) using collagen, botulinum toxin, or other wrinkle treatments
    * Within 6 months before Visit 1 (screening) undergoing invasive laser, deep dermabrasion, or other procedures or surgeries related to wrinkle treatment in the eye area
    * Insertion of permanent skin expansion implants like Softform or silicone in the eye area before screening
    * Starting or receiving a new oral or topical anti-wrinkle medication with wrinkle prevention effects within 3 months before Visit 1 (screening)
12. Individuals who have undergone the following drug therapies that could affect the evaluation of the investigational medical device:

    * Use of NSAIDs, antiplatelet agents, anticoagulants, immunosuppressants within 2 weeks before Visit 1 (screening), or required during the clinical trial period (excluding low-dose aspirin (100 mg, up to 300 mg/day))
    * Use of topical agents (steroids, retinoids: only medications, not cosmetics) in the eye area within 1 month before Visit 1 (screening) or planned use during the clinical trial
13. Individuals who have received a COVID-19 vaccine within 3 weeks before the application of the investigational medical device or are planned to receive it within 4 weeks after application
14. Individuals with ongoing infectious diseases, including COVID-19, or suspected COVID-19 infection within 2 weeks before screening
15. Individuals who have been administered or undergone other investigational drugs or devices within 1 month before Visit 1 (screening), or within 6 months for studies related to crow's feet wrinkles
16. Individuals with positive results for viral tests (HBs Ag, HCV Ab, HIV Ab) performed at Visit 1 (screening) or within 1 month before screening
17. Individuals with a history of alcohol or drug addiction
18. Pregnant or breastfeeding women
19. Individuals planning to become pregnant during the clinical trial or those who, along with their partners (or spouses), do not agree to use medically acceptable contraception methods (examples include: hormonal contraceptives, proven failure rates intrauterine devices (IUDs), double barrier methods, sterilization)
20. Individuals deemed unsuitable for participation in the clinical trial based on the investigator's judgment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2025-11-27 (Actual)

PRIMARY OUTCOMES:
Improvement rate of IGA-LCL wrinkle severity by external independent evaluators | 18 weeks
  Improvement rate of 1 point or more on the crow's feet at rest IGA-LCL severity scale by external independent evaluators at 18 weeks after initial injection

SECONDARY OUTCOMES:
Improvement rate of IGA-LCL wrinkle severity by external independent evaluators | 8, 10 weeks
  Improvement rate of 1 point or more on the crow's feet at rest IGA-LCL severity scale by external independent evaluators at 8, 10 weeks after initial injection
Change in GAIS scores assessed by an independent evaluator | 8, 10, 18 weeks
  Change in GAIS scores assessed by an independent evaluator at 8, 10, 18 weeks after initial injection
Improvement rate of GAIS for both crow's feet as assessed by an independent evaluator | 8, 10, 18 weeks
  Improvement rate of GAIS for both crow's feet as assessed by an independent evaluator at 8, 10, 18 weeks after initial injection
Change in GAIS scores assessed by the subject | 8, 10, 18 weeks
  Change in GAIS scores assessed by the subject at 8, 10, 18 weeks after initial injection
Improvement rate of GAIS for both crow's feet as assessed by the subject | 8, 10, 18 weeks
  Improvement rate of GAIS for both crow's feet as assessed by the subject at 8, 10, 18 weeks after initial injection

CONTACTS AND LOCATIONS:
Overall Officials: Beom Joon Kim, M.D., Study Director — Dermatology
Locations (1):
- Chung-Ang University Hospital, Seoul, Heukseok-ro, Dongjak-gu, South Korea

IPD SHARING:
Plan to Share IPD: No